CLINICAL TRIAL: NCT03184714
Title: The Effectiveness of Noninvasive Positive Pressure Ventilation Treatment in Overlap Syndrome
Brief Title: Noninvasive Positive Pressure Ventilation in Overlap Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1304403B
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; Sleep Apnea Syndromes; Non-invasive Positive Pressure Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: non-invasive positive pressure ventilation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Interventional group (Experimental): NIPPV as treatment of OS
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: NIPPV — BiPAP treatment for 3 years
  Arms: Interventional group

SUMMARY:
Chronic obstructive pulmonary diseases (COPD) coexisting with obstructive sleep apnea is called overlap syndrome (OS). Patients with OS seem to have worse prognosis than patients with only one disorder. Noninvasive positive pressure ventilation is an efficient treatment in obstructive sleep apnea, but the effectiveness in improving outcomes of OS patients is still not fully investigated. The aim of this non-randomized concurrent control trial is to evaluate noninvasive positive pressure ventilation's effectiveness in OS patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD and sleep apnea dyspnea syndrome

Exclusion Criteria:

* patients with non-stable hemodynamics;
* patients with limited life expectancy;
* patients with other severe respiratory diseases;
* patients with motor neuron diseases;
* patients with contraindications for NIPPV

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD acute exacerbations | 3 years
  total times of COPD acute exacerbations

SECONDARY OUTCOMES:
COPD assessment test (CAT) score | 3 years
  symptom score of COPD
modified British medical research council (mMRC) score | 3 years
  dyspnea score
all-cause mortality | 3 years
  survival rate in %

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided